CLINICAL TRIAL: NCT06548945
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-escalation Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics (PK/PD) of a Single Dose of GZR18 Injection in Obese/Overweight Subjects
Brief Title: A Phase I Study of GZR18 Injection in Obese/Overweight Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GL-GLP-CH1017
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR18 (Experimental)
  Interventions: Drug: GZR18
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GZR18 — 5 mg-maximum tolerated dose (MTD), single dose
  Arms: GZR18
Other: Placebo — administered the same volume as GZR18
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-escalation phase I clinical study. A sequential design is used in this trial with a single dose escalation climb test, to investigate the safety, tolerability, and PK/PD characteristics of GZR18 injection in Chinese obese/overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects sign the informed consent form (ICF) voluntarily.
* Chinese adult subjects, both male and female.
* 18 to 65 years old (including both ends) at screening.
* BMI≥26.0 kg/m2 at screening.
* Stable weight before screening (i.e. self-reported weight change less than 5 kg within 8 weeks before screening).
* Female subjects have negative serum Human Chorionic Gonadotropin (HCG) during screening and baseline periods.
* Subjects have good daily habits and can maintain good communication with investigators and comply with various requirements of clinical trials.

Exclusion Criteria:

* Lactating women.
* History of fainting with blood and needles.
* Known or suspected allergy to study related products; or drug/food allergy history; or allergy-related diseases history.
* Subjects who have participated in other clinical trials and given investigational drugs or medical device interventions within 90 days before screening.
* History of drug abuse within 1 year before screening, or positive results in drug abuse screening (urine).
* Smokers who smoke ≥ 5 cigarettes per day within the previous 3 months before screening or cannot refrain from smoking throughout the trial period.
* Any vaccine has been used within 28 days before administration, as well as any vaccine that may be used throughout the trial period.
* Other scenarios judged by the investigator to render the subjects unsuitable for participating in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
TEAE | 50 days
  Incidence of Treatment Emergent Adverse Event(s)
Anti-Drug Antibody (ADA) and Neutralizing Antibody (Nab) | 50 days

SECONDARY OUTCOMES:
Cmax | 50 days
  Maximum plasma drug concentration
AUClast | 50 days
  area under the curve from 0 through the time of the last accurately measurable concentration
AUC0-inf | 50 days
  area under the curve extrapolated to infinity
Tmax | 50 days
  time to maximum plasma drug concentration
λz | 50 days
  elimination rate constant
t1/2 | 50 days
  half-life
tlag | 50 days
  lag time
CL/F | 50 days
  apparent clearance
Vz/F | 50 days
  volume of distribution/F
AUC%extra | 50 days
  percent of AUC0-inf extrapolated
MRT | 50 days
  mean residence time
Weight | 50 days
Body Mass Index (BMI) | 50 days

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Zhao, Ph.D, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Gan & Lee Pharmaceuticals Co., Ltd, Beijing, China